CLINICAL TRIAL: NCT05673148
Title: A Pragmatic Randomized Phase III Trial Evaluating Total Ablative Therapy for Patients With Limited Metastatic Colorectal Cancer: Evaluating Radiation, Ablation, and Surgery (ERASur)
Brief Title: Testing the Addition of Total Ablative Therapy to Usual Systemic Therapy Treatment for Limited Metastatic Colorectal Cancer, The ERASur Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A022101; NCI-2022-09253 (Other: NCI)
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (TAT, SOC chemotherapy (Experimental): Patients undergo TAT on study, consisting of SABR with or without surgical resection and/or microwave ablation. Patients also receive SOC chemotherapy on study. Patients also undergo CT or MRI or PET/CT scans throughout the trial.
  Interventions: Procedure: Stereotactic Ablative Radiotherapy; Procedure: Resection; Procedure: Microwave Ablation; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Arm 2 (SOC chemotherapy) (Active Comparator): Patients receive SOC chemotherapy on study. Patients also undergo Patients also undergo CT or MRI or PET/CT scans throughout the trial.
  Interventions: Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Stereotactic Ablative Radiotherapy — Undergo SABR
  Other Names: SABER; SABR/SBRT
  Arms: Arm 1 (TAT, SOC chemotherapy
Procedure: Resection — undergo surgical resection
  Other Names: Surgical resection
  Arms: Arm 1 (TAT, SOC chemotherapy
Procedure: Microwave Ablation — undergo microwave ablation
  Other Names: Ablation
  Arms: Arm 1 (TAT, SOC chemotherapy
Drug: Chemotherapy — Receive SOC chemotherapy
  Other Names: Chemo
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan

SUMMARY:
This phase III trial compares total ablative therapy and usual systemic therapy to usual systemic therapy alone in treating patients with colorectal cancer that has spread to up to 4 body sites (limited metastatic). The usual approach for patients who are not participating in a study is treatment with intravenous (IV) (through a vein) and/or oral medications (systemic therapy) to help stop the cancer sites from getting larger and the spread of the cancer to additional body sites. Ablative means that the intention of the local treatment is to eliminate the cancer at that metastatic site. The ablative local therapy will consist of very focused, intensive radiotherapy called stereotactic ablative radiotherapy (SABR) with or without surgical resection and/or microwave ablation, which is a procedure where a needle is temporarily inserted in the tumor and heat is used to destroy the cancer cells. SABR, surgical resection, and microwave ablation have been tested for safety, but it is not scientifically proven that the addition of these treatments are beneficial for your stage of cancer. The addition of ablative local therapy to all known metastatic sites to the usual approach of systemic therapy could shrink or remove the tumor(s) or prevent the tumor(s) from returning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate and compare overall survival (OS) (measured from time of randomization) in patients with newly diagnosed oligometastatic colorectal cancer (oCRC) treated with total ablative therapy (TAT) in addition to standard of care (SOC) systemic therapy versus SOC systemic therapy.

SECONDARY OBJECTIVES:

I. To evaluate and compare event-free survival (EFS) (measured from time of randomization) between the two treatment arms.

II. To assess the adverse events (AE) profile within each of the two treatment arms.

III. To evaluate the time to local recurrence (TLR) (measured from completion of TAT) in patients with newly diagnosed oCRC treated with TAT + SOC systemic therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients undergo TAT on study, consisting of SABR with or without surgical resection and/or microwave ablation. Patients also receive SOC chemotherapy on study. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) or positron emission tomography (PET)/CT scans throughout the trial.

ARM 2: Patients receive SOC chemotherapy on study. Patients also undergo Patients also undergo CT or MRI or PET/CT scans throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION (STEP 0): Histologically-confirmed metastatic colorectal adenocarcinoma
* PRE-REGISTRATION (STEP 0): No known microsatellite instable (MSI) tumor
* PRE-REGISTRATION (STEP 0): No known BRAF V600E mutation
* PRE-REGISTRATION (STEP 0): Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. No known peritoneal and/or omental metastases. If radiologic studies suggest the presence of peritoneal disease, a diagnostic laparoscopy is recommended to verify the absence of peritoneal implants
* PRE-REGISTRATION (STEP 0): Primary tumor is already resected OR primary tumor is surgically amenable to resection, as determined by consultation and documentation with surgeon or documentation of discussion in the institutional multi-disciplinary tumor board where a surgeon confirms resectability. Patients with unresectable primary tumors are not eligible
* PRE-REGISTRATION (STEP 0): Four (4) or fewer apparent sites of metastatic disease based on review by local medical team of baseline radiographic imaging obtained prior to initiation of systemic therapy.

  * Sites of metastatic disease must be radiographically evident, but pathologic confirmation is not required.
  * Liver-only metastatic disease is NOT permitted. For patients with liver metastases, there must be at least one other site of metastasis in addition to the liver to be eligible for this study.
  * Metastatic lesions must be amenable to any combination of surgical resection, microwave ablation, and/or stereotactic ablative body radiation therapy (SABR). SABR is required for at least one lesion. Therefore, the patient must be seen by a radiation oncologist in consultation to verify eligibility.
  * Single sites include:

    * Each hemiliver (right and left), each lobe of the lungs, each adrenal gland, lymph nodes amenable to a single resection or treatment in a single SABR field, bone metastases amenable to treatment in a single SABR field
* PRE-REGISTRATION (STEP 0): Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* PRE-REGISTRATION (STEP 0): A maximum of 16 weeks (4 months) of systemic therapy may be administered prior to pre-registration
* REGISTRATION (STEP 1): Patients must have no overt evidence of disease progression during systemic therapy prior to registration
* REGISTRATION (STEP 1): Not eligible for hepatic artery infusion pump (HAIP) therapy or benefit of HAIP therapy is undefined
* REGISTRATION (STEP 1): Patients must have measurable disease per RECIST v1.1
* REGISTRATION (STEP 1): Patients must be receiving (or have received) first-line systemic therapy for metastatic disease for a minimum of 16 weeks (4 months) and a maximum of 24 weeks (6 months)
* REGISTRATION (STEP 1): Prior definitive therapy, including adjuvant chemotherapy, must have been completed at least 12 months prior to diagnosis of metastatic disease
* REGISTRATION (STEP 1): Not pregnant and not nursing, because this study involves an agent or treatment that has known genotoxic, mutagenic, and teratogenic effects.

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 14 days prior to registration is required
* REGISTRATION (STEP 1): Age >= 18 years
* REGISTRATION (STEP 1): Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
* REGISTRATION (STEP 1): Absolute neutrophil count (ANC) >= 1,500/mm^3
* REGISTRATION (STEP 1): Platelet count >= 50,000/mm^3
* REGISTRATION (STEP 1): Creatinine =< 1.5 x upper limit of normal (ULN) OR calculated (calc.) creatinine clearance >= 30 mL/min

  * Calculated using the Cockcroft-Gault equation
* REGISTRATION (STEP 1): Total bilirubin =< 1.5 x ULN
* REGISTRATION (STEP 1): Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x ULN

  * In the event of metastatic liver disease, =< 5 x ULN
* REGISTRATION (STEP 1): Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Note: HIV testing is not required for eligibility
* REGISTRATION (STEP 1): No other planned concurrent investigational agents while on study

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2028-07-03 (Estimated); Study Completion 2032-08-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of randomization to the date of death due to all causes, assessed up to 5 years
  o Description: The hazard ratio (HR) for OS will be estimated using a stratified Cox proportional hazards model and the 95% confidence interval (CI) for the HR will be provided. The Kaplan-Meier methodology will be used to estimate the median OS for each treatment arm, and Kaplan-Meier curves will be produced. OS will also be compared between treatment arms using the log rank test

SECONDARY OUTCOMES:
Event Free Survival (EFS) | From randomization to the date of first documented progression, recurrence, or death due to all causes, whichever occurs first, assessed up to 5 years
  The hazard ratio (HR) for EFS will be estimated using a stratified Cox proportional hazards model and the 95% confidence interval (CI) for the HR will be provided. The Kaplan-Meier methodology will be used to estimate the median EFS for each treatment arm, and Kaplan-Meier curves will be produced. EFS will also be compared between treatment arms using the log rank test.
• Incidence of Adverse Events (AEs), assessed using National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0 (v5.0) | Up to 5 years
  Defined as the proportion of patients experienced at least one Grade 3, Grade 4, or Grade 5 of each type of AE. The maximum grade for each type of adverse events that are possibly, probably, or definitely related to study treatments will be recorded for each patient. The frequency tables will be reviewed to determine the patterns. The overall adverse event rates for grade 3 or higher adverse events will be compared between two treatment groups using Chi-square test (or Fisher's exact test if the data in the contingency table is sparse).
Time to local recurrence (TLR) | from the end of TAT to the date of first documented recurrence at any disease site treated with TAT, assessed up to 5 years after randomization
  TLR will be measured only for patients who receive treatment with TAT and is defined as the time from the end of TAT until the date of first documented recurrence at any disease site treated with TAT. The Kaplan-Meier methodology will be used to estimate the median TLR for patients treated with TAT , and a Kaplan-Meier curve will be produced.

CONTACTS AND LOCATIONS:
Locations (182):
- United States (182):
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - University of Illinois, Chicago, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Northwell Health Physicians Partners Radiation Medicine at Queens, Forest Hills, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Queens Cancer Center, Rego Park, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Westchester Medical Center, Valhalla, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Valley Medical Center, Renton, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hitchcock KE, Miller ED, Shi Q, Dixon JG, Gholami S, White SB, Wu C, Goulet CC, George M, Jee KW, Wright CL, Yaeger R, Shergill A, Hong TS, George TJ, O'Reilly EM, Meyerhardt JA, Romesser PB. Alliance for clinical trials in Oncology (Alliance) trial A022101/NRG-GI009: a pragmatic randomized phase III trial evaluating total ablative therapy for patients with limited metastatic colorectal cancer: evaluating radiation, ablation, and surgery (ERASur). BMC Cancer. 2024 Feb 13;24(1):201. doi: 10.1186/s12885-024-11899-2. PMID 38350888
- [Derived] Miller ED, Hitchcock KE, Romesser PB. Oligometastatic Colorectal Cancer: A Review of Definitions and Patient Selection for Local Therapies. J Gastrointest Cancer. 2023 Dec;54(4):1116-1127. doi: 10.1007/s12029-022-00900-5. Epub 2023 Jan 18. PMID 36652155